CLINICAL TRIAL: NCT03924622
Title: Prevention of Pressure Injuries During Aeromedical Evacuation or Prolonged Field Care
Brief Title: Pressure Injury Prevention in AE and PFC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue to conduct study procedures due to pandemic
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Elizabeth Bridges, Professor, School of Nursing: Dept: Biobehavioral Nursing and Health Informatics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00006022
Record Dates: First submitted 2019-04-10; First posted 2019-04-23 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-03

CONDITIONS: Pressure Injury; Military Activity
Keywords: Pressure injury/prevention; Military Nursing; Risk Reduction
MeSH Terms: conditions — Pressure Ulcer; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Stratified randomized control trial with subjects assigned to either the simulated aeromedical evacuation (standard mattress or vacuum spine board) or Prolonged Field Care arms with or without the intervention. Stratification will be based on body fat percentage. Study does not involve FDA-regulated drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: Mepilex on Litter + AE Mattress + 30 degree backrest (Experimental): Intervention: Mepilex
  Interventions: Device: Mepilex
- Group 2: Without Mepilex on Litter + AE mattress + backrest (No Intervention): Intervention: Control (no Mepilex)
- Group 3: Mepilex on VSB on AE mattress (Experimental): Intervention: Mepilex
  Interventions: Device: Mepilex
- Group 4: Without Mepilex on VSB on AE mattress (No Intervention): Intervention: Control (no Mepilex)
- Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon litter (Experimental): Intervention: LiquiCell mat
  Interventions: Device: LiquiCell
- Group 6: PFC Without LiquiCell on Talon Litter (No Intervention): Intervention: Control (no LiquiCell)

INTERVENTIONS:
Device: Mepilex — Mepilex Border Sacrum dressing is a multi-layered soft silicone dressing that is a recommended strategy to augment standard nursing interventions (i.e., repositioning, offloading) to prevent pressure injuries. The dressing will be placed on the sacrum.
  Arms: Group 1: Mepilex on Litter + AE Mattress + 30 degree backrest; Group 3: Mepilex on VSB on AE mattress
Device: LiquiCell — LiquiCell is a thin layer of low-viscosity fluid contained in a series of bursa-like pouches. Baffles within each pouch channel the liquid to disperse pressure and the volume of liquid in the pouch is so small that there is no pressure-build up. LiquiCell is available commercially as a 36 X 18-inch mattress overlay (LiquiCell Shear Reducing Mattress Overlay) with a soft pliable top and a non-slip bottom. The overlay is positioned from the shoulders to below the hips to minimize shear.
  Arms: Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon litter

SUMMARY:
This study evaluates the effect of a multilayer skin dressing (Mepilex) placed on the sacrum or a fluid filled pad (LiquiCell) on risk factors for pressure injuries under conditions consistent with military long-distance transport or prolonged field care. Participants will be assigned to one of six groups - air transport, air transport on a spinal immobilization surface with or without Mepilex or on a field stretcher with or without LiquiCell.

DETAILED DESCRIPTION:
Combat casualties undergoing long distance aeromedical evacuation (AE), particularly casualties who are immobilized because of possible spine injuries, and casualties who required prolonged field care are at increased risk for pressure injuries. The risk factors pressure and shear are potentially modifiable via solutions appropriate for these austere conditions. Two interventions (Mepilex and LiquiCell) will be evaluated under conditions simulating military medical transport on a standard stretcher or with spinal immobilization in a vacuum spine board (VSB) or on a military stretcher used under field conditions. Mepilex is a multi-layer dressing that can be placed on the skin (sacrum/buttocks) and LiquiCell is a pad filled with pockets of fluid that is placed under the back and buttocks. The effect of these interventions compared to not using them will be studied under the three conditions with or without the intervention (Mepilex or LiquiCell) using measures obtained on the lower back/sacrum including skin interface pressure, oxygen, moisture, and temperature and a cytokine indicating possible tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18 to 55
* Meet the physical standards for military personnel
* Weigh less than 250 pounds
* Be able to remain in the study position for the duration of the study.

Exclusion Criteria

* Previous injuries to sacrum/buttocks with scarring
* History of pressure injuries
* Cardiovascular disease
* Neurological disease that would affect vascular response
* Diabetes
* History of malignancy
* Current skin condition (e.g., eczema or psoriasis)
* Current neck/back pain or history of chronic neck/back pain
* Known vertebral/spinal cord disease/injury (scoliosis, kyphosis, or lordosis)
* Self-reported pregnancy
* Concern about ability to remain in the vacuum spine board for 120 minutes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bridges, PhD, RN, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bridges E, Whitney JD, Burr R, Tolentino E. Reducing the Risk for Pressure Injury During Combat Evacuation. Crit Care Nurse. 2018 Apr;38(2):38-45. doi: 10.4037/ccn2018223. PMID 29606674

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest; Group 3: Mepilex on VSB on WELP Mattress: Intervention: Mepilex
  Mepilex: Mepilex Border Sacrum dressing is a multi-layered soft silicone dressing that is a recommended strategy to augment standard nursing interventions (i.e., repositioning, offloading) to prevent pressure injuries. The dressing will be placed on the sacrum.
- Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest; Group 4: Without Mepilex on VSB on WELP Mattress: Intervention: Control (no Mepilex)
Period: Overall Study
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Started | 12 | 12 | 12 | 12 | 12 | 12
Completed | 10 | 9 | 9 | 8 | 9 | 9
Not Completed | 2 | 3 | 3 | 4 | 3 | 3
Not completed — Study closed due to pandemic with approval of funding agency/IRB | 2 | 3 | 3 | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All individuals with baseline data
Groups:
- Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest: Intervention: Mepilex Study surface Litter + WELP mattress pad with 30 degree backrest.
  Mepilex: Mepilex Border Sacrum dressing is a multi-layered soft silicone dressing that is a recommended strategy to augment standard nursing interventions (i.e., repositioning, offloading) to prevent pressure injuries. The dressing will be placed on the sacrum.
- Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest: Intervention: Control (no Mepilex)
  Study surface Litter + WELP mattress pad with 30 degree backrest. No Mepilex
- Group 3: Mepilex on VSB on WELP Mattress: Intervention: Mepilex Litter + WELP mattress + Vacuum Spineboard.
  Mepilex: Mepilex Border Sacrum dressing is a multi-layered soft silicone dressing that is a recommended strategy to augment standard nursing interventions (i.e., repositioning, offloading) to prevent pressure injuries. The dressing will be placed on the sacrum.
- Group 4: Without Mepilex on VSB on WELP Mattress: Intervention: Control (no Mepilex)
  Litter + WELP mattress + Vacuum Spineboard. No Mepilex
- Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter: Intervention: LiquiCell mat Talon litter LiquiCell: LiquiCell is a thin layer of low-viscosity fluid contained in a series of bursa-like pouches. Baffles within each pouch channel the liquid to disperse pressure and the volume of liquid in the pouch is so small that there is no pressure-build up. LiquiCell is available commercially as a 36 X 18-inch mattress overlay (LiquiCell Shear Reducing Mattress Overlay) with a soft pliable top and a non-slip bottom. The overlay is positioned from the shoulders to below the hips to minimize shear.
- Group 6: PFC Without LiquiCell on Talon Litter: Intervention: Control (no LiquiCell)
  Talon litter
- Total: Total of all reporting groups
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter | Total
Number analyzed (Participants) | 10 | 9 | 9 | 8 | 9 | 9 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (10.6) | 26.7 (7.3) | 25.3 (12.3) | 24.8 (5.9) | 23.9 (8.8) | 25 (8) | 29 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 6 | 6 | 6 | 8 | 40
  Male | 2 | 3 | 3 | 2 | 3 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 8 | 9 | 8 | 9 | 9 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 5 | 5 | 4 | 4 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 6 | 3 | 3 | 2 | 5 | 5 | 24
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 2
Body Fat Percent [Mean (Standard Deviation); unit: Percent body fat] | 29 (10.6) | 26.7 (7.3) | 25.3 (12.3) | 24.8 (5.9) | 23.9 (8.8) | 25.0 (8.0) | 25.8 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin-1/Total Protein (Skin)
Description: Skin cytokine (IL-1) and total protein will be obtained using a small strip of specialized tape placed on the sacrum/buttocks. After 1-minute application the tape is removed and analyzed for quantity of interleukin-1 (indicator of skin irritation)
Time Frame: Baseline through study completion - approximately 120 minutes
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Number analyzed (Participants) | 10 | 9 | 9 | 8 | 9 | 9
Ratio | -1.9 (2.7) | -0.8 (2.7) | 0.13 (2.4) | -4 (2.2) | -3.5 (2.7) | 0.14 (0.3)

2. Primary Outcome: Change in Transcutaneous Tissue Oxygen (TcPO2)
Description: Tissue oxygen is measured continuously on the sacrum using a noninvasive sensor and on the midsternum (midchest) as a control
Time Frame: Measured continuously during the baseline (sidelying), supine (120 minutes) and post-sidelying (15 minutes) periods
Population: All subjects exposed to condition. Data collection stopped at 60 minutes due to critically low TcPO2 - Group 2 (n = 1); Group 5 (n = 5), Group 6 (n =5). One subject (Group 6) all data collection stopped at 90 minutes due to general discomfort. Complete data analysis for all subjects through 60 minutes. Complete (120 minutes of data available Gp 1 = 10; Gp 2 = 8, Gp 3 = 9; Gp 4 = 8; Gp 5 = 4; Gp 6 = 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Number analyzed (Participants) | 10 | 8 | 9 | 8 | 4 | 3
mm Hg | -15 (26) | -25 (25) | -4 (23) | -6 (16) | -54 (24) | -53 (17)

3. Primary Outcome: Change in Skin Moisture (Epidermal and Subepidermal)
Description: Two components of skin moisture will be measured on the sacrum using the Delfin MoistureMeter. The epidermal moisture, which reflects perspiration and subepidermal moisture , which reflects water content of the tissues. The values range from 1-80, with higher numbers reflecting increased moisture.
Time Frame: Baseline (before lying down) and after 120 minutes supine
Population: All participants exposed to the condition
Measure: Mean (Standard Deviation); unit: Tissue Dielectric Constant (TDC)
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Number analyzed (Participants) | 10 | 9 | 9 | 8 | 9 | 9
Tissue Dielectric Constant (TDC) | 1.5 (2) | 2 (3.8) | 1.1 (2.2) | 2.1 (2.8) | -0.1 (2) | 0.1 (1.3)

4. Primary Outcome: Change in Skin Temperature
Description: Skin temperature will be measured continuously on the sacrum using a laser doppler probe.
Time Frame: Measured continuously during the baseline (sidelying), supine (120 minutes) and post-sidelying (15 minutes) periods
Population: All participants exposed to the condition
Measure: Mean (Standard Deviation); unit: Degrees centigrade
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Number analyzed (Participants) | 10 | 9 | 9 | 8 | 9 | 9
Degrees centigrade | 3.8 (1.3) | 3.1 (1) | 3.7 (0.8) | 3.2 (1) | 2 (2) | 1.1 (0.9)

5. Primary Outcome: Change in Skin Interface Pressure
Description: The pressure between the support surface and the skin will be measured continuously during the supine position using the X Sensor system. This system measures force/unit area (e.g., pressure). The peak and average pressure on the sacrum/buttocks will be measured.
Time Frame: Continuously during the supine phase of the study (120 minutes)
Population: All participants exposed to the condition
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Number analyzed (Participants) | 10 | 9 | 9 | 8 | 9 | 9
mm Hg | 46 (8) | 52 (10) | 52 (10) | 66 (22) | 66 (27) | 78 (47)

6. Secondary Outcome: Change in Pressure-Discomfort (Category Partitioning Scale-50)
Description: This scale asks the participant to describe in verbal terms the pressure intensity or discomfort associated with the stimulus (i.e., sacral/buttocks pressure or discomfort). The participant can then fine tune their assessment using a numeric score. The final score is an analog. The score ranges from 0-52, with higher scores indicating higher pressure or more severe discomfort. The investigator will ask the participant to limit their evaluation to the pressure/discomfort sensed on the sacrum/buttocks, but the investigator will also ask the participants to identify on their body where they are experiencing the most pressure/discomfort.
Time Frame: The score will be obtained at baseline and every 30 minutes in the supine position (total 5 measurements).
Population: All participants exposed to the condition
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
Number analyzed (Participants) | 10 | 9 | 9 | 8 | 9 | 9
Scores on a scale | 7.7 (8.1) | 8 (10.4) | 9.1 (7.3) | 5.4 (4.2) | 8.7 (13.4) | 12.3 (11.1)

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | Group 1: Mepilex on Litter + WELP Mattress + 30 Degree Backrest | Group 2: Without Mepilex on Litter + WELP Mattress +30 Degree Backrest | Group 3: Mepilex on VSB on WELP Mattress | Group 4: Without Mepilex on VSB on WELP Mattress | Group 5 Prolonged Field Care (PFC) - LiquiCell on Talon Litter | Group 6: PFC Without LiquiCell on Talon Litter
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03924622/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03924622/SAP_001.pdf